CLINICAL TRIAL: NCT06159712
Title: Comparative Study of High-Efficacy Disease Modifying Treatment of Relapsing Multiple Sclerosis
Acronym: CoSHEDRMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Gødstrup Hospital (Other); Regionshospitalet Viborg, Skive (Other); Sorbonne University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CoSHED
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Researchers compare immunologic, virologic and epigenetic factors in patients with multiple sclerosis in standard 2.line treatment with ocrelizumab, rituximab, ofatumumab and natalizumab by taking extra blood samples and compare it to a healthy control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Ocrelizumab (Other): Patients with active multiple sclerosis starting standard treatment with ocrelizumab
  Interventions: Other: Blood samples
- Rituximab (Other): Patients with active multiple sclerosis starting standard treatment with rituximab
  Interventions: Other: Blood samples
- Ofatumumab (Other): Patients with active multiple sclerosis starting standard treatment with ofatumumab
  Interventions: Other: Blood samples
- Natalizumab (Other): Patients with active multiple sclerosis starting standard treatment with natalizumab
  Interventions: Other: Blood samples
- Healthy controls (Other): An age and gender matched healthy control group
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Extra blood samples

SUMMARY:
The goal of this prospective, multi-center, non-blinded, non-randomized, non-intervention clinical trial is to compare immunologic, virologic and epigenetic factors in patients with active multiple sclerosis in standard 2.line treatment with ocrelizumab, rituximab, ofatumumab or natalizumab in Region Midt, Denmark. It aims to answer how the immunologic, virologic and epigenetic response in these patients are compared to healthy controls, and analyze their treatment effect in relation to this response. Participants will get an extra blood sample, when they have their routine blood samples taken.

DETAILED DESCRIPTION:
The CoSHED RMS study will include patients with active multiple sclerosis aged 18-65 years fulfilling the criteria for 2. line treatment and starting treatment with one of the four high-efficacy disease modifying treatments ocrelizumab, rituximab, ofatumumab or natalizumab. Researchers will compare immunologic, virologic and epigenetic parameters in the four treatment groups to a age and gender matched healthy control group. The study duration is 12 months, and patients can continue in an extension phase for additional 12 month. The primary endpoint is changes in B cell populations between the four treatments within 12 months. The study will evaluate a number of efficacy and safety endpoints using clinical, MRI, routine blood samples and research biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis diagnosis and definition of disease course according to the 2017 McDonald criteria
* Expanded disability status scale (EDSS) ≤6.5
* Signed written informed consent
* Fulfilling criteria for active MS: Treatment naïve relapsing remitting multiple sclerosis (RRMS) patients (never treated, or no DMT the previous 2 years):

  * 2 relapse previous 12 months OR

    1 relapse previous 12 months with severe residual symptoms and EDSS ≥ 3.0 OR

    1 relapse previous 12 months AND ≥9 T2 lesions on brain and/or spinal cord MRI AND
    1. contrast-enhancing lesion or ≥1 new or enlarging T2 lesion on brain and/or spinal cord MRI previous 12 month

       Previously treated RRMS patients:
  * 1 relapse previous 12 months OR
  * 1 contrast-enhancing lesion or ≥2 new/enlarging T2 lesions on brain and/or spinal cord MRI previous 12 months

Exclusion Criteria:

* Pregnancy or breast feeding
* Lack of effective contraception for women of child-bearing potential (effective contraception include oral contraception, intrauterine devices and other forms of contraception with failure rate <1%)
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to randomization
* Known active malignant disease
* Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Positive test for HIV, hepatitis B or C, or tuberculosis
* Negative test for varicella zoster
* Lymphopenia grade 2 (0.5 to 0.8 × 10^9/L) or higher grades of lymphopenia (in case of switching from fingolimod lymphopenia grade 2 can be accepted if lymphocytes are rising markedly compared to on treatment levels)
* Neutropenia grade 2 (1.0 to 1.5 × 10^9/L) or higher grades
* Thrombocytopenia grade 2 (50 to 75 × 10^9/L) or higher grades
* Previous treatment with alemtuzumab or hematopoietic stem-cell transplantation
* Previous treatment with cladribine, CD20-depleting antibodies, daclizumab or other immune suppressive treatment which is judged to still exert immune suppressive effect by treating physician
* Methylprednisolone treatment within 1 month of baseline visit
* Findings on the screening MRI judged to preclude participation by the treating physician
* Other diseases judged to be relevant by the treating physician
* Contraindication to MRI
* Known allergy or hypersensitivity to rituximab or ocrelizumab, rituximab, ofatumumab or natalizumab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in B cell populations | 1 year
  Changes in B cell populations in the four treatment groups

OTHER OUTCOMES:
Relapses | 1 year
  Number of patients with relapse or relapses from start of treatment from baseline to 12 months
Annualized Relapse Rate | 1 year
  Annualized Relapse Rate based on the total amount of relapses per year from baseline to 12 months
T-cells, B-cell subsets and monocyte-subsets | 1 year
  Changes in frequency of T-cells, B-cell-subsets and monocyte-subsets from baseline, 6 months and to 12 months
EBV | 1 year
  Changes in Epstein Barr-Virus DNA load from baseline, 6 months and to 12 months
HERVs | 1 year
  Changes in Human Endogenous Retrovirus expression from baseline, 6 months and to 12 months
Complement | 1 year
  Changes in complement system activity from baseline, 6 months and to 12 months
MRI lesions | 1 year
  Changes in number of lesions on MRI scans of the brain from baseline, 6 months and to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Morten Stilund, MD, Study Director — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: After finishing the study, available for 1 year